CLINICAL TRIAL: NCT03731975
Title: Efficacy of Endodontic Treatment Using CTZ Paste in Primary Teeth: Randomized Clinical Trial
Brief Title: Endodontic Treatment Using CTZ Paste in Primary Teeth
Acronym: SLM2204
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, Principal Investigator, Clinical Professor, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SLM4
Record Dates: First submitted 2018-10-25; First posted 2018-11-06 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Pulpectomy Agents
Keywords: Tooth, deciduous; Pulp Capping and Pulpectomy Agents; Pulpectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTZ Paste (Active Comparator): Endodontic treatment with CTZ paste.
  Interventions: Procedure: CTZ Paste
- GP Paste (Experimental): Endodontic treatment with Guedes-Pinto paste.
  Interventions: Procedure: GP Paste

INTERVENTIONS:
Procedure: CTZ Paste — Tooth allocated to this group will be treated with CTZ paste, according to the Cappielo's protocol (1964), updated by Moura et al. (2016).
  Arms: CTZ Paste
Procedure: GP Paste — Tooth allocated to this group will be treated with Guedes-Pinto paste, according to the Guedes-Pinto's protocol (1981), updated by Mello-Moura et al. (2011).
  Arms: GP Paste

SUMMARY:
The aim of this study is to evaluate the efficacy of CTZ Paste in primary teeth, compared to endodontic treatment with Guedes-Pinto Paste. This is a multicenter, randomized, double-blind (patient), controlled and non-inferiority clinical study on 174 primary molars and 174 primary incisors of 3-6 years-old children with carious lesions with pulp involvement. The sample unit will be the tooth, which will be randomized into two groups. The teeth allocated to the experimental group will be treated with CTZ Paste, whereas the treatment of those teeth allocated to the control group will employ the Guedes-Pinto Paste. The procedures performed will be evaluated clinically and radiographically at 6 and 12 months. Secondary outcomes such as cost, discomfort, satisfaction and quality of life will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 3 to 6 years and 11 months;
* children present at least one upper or lower molar or primary upper incisor with untreated carious lesion with pulp envelopment;
* children assent to participate in the study through collaborative behavior;
* children's parents/guardians consent to their participation by signing the Informed Consent Form (ICF).

Exclusion Criteria:

* tooth with carious lesion involving three or more dental surfaces, making the restoration extremely difficult or impossible;
* tooth with internal or external resorption in more than 1/3 of the root length;
* tooth whose crypt of the successor permanent is affected;
* tooth which have less than 2/3 of the root;
* patients who present health problems with oral impairment.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical and radiographical efficacy of the endodontic treatment | 12 Months
  The tooth will be evaluated according to the presence of mobility (yes or no) and regarding radiolucency area on initial and final radiography (measured and compared with the program ImageJ).

SECONDARY OUTCOMES:
Cost-efficacy | Through study completion (12 months)
  The costs of each treatment procedure will be calculated and compared with thresholds values for intervention cost-effectiveness by region, determined by World Health Organization (http://www.who.int/choice/costs/CER_levels/en/). These values will be combined with the evaluated efficacy of the treatments (according description of Outcome 1).
Children's satisfaction with treatment | Through study completion (12 months)
  The satisfaction of each treatment will be evaluated using the Wong-Baker Facial Scale (Wong & Baker, 1988). The patient will be asked to choose the face that is more similar to how he/she felt during the treatment. The answer should be given solely by the child, which means no parental or professional interferences.
Parents/Guardians' satisfaction with children's treatment | Through study completion (12 months)
  The parents' satisfaction with each treatment will be evaluated using the Parent's Questionnaire about Teeth Appearance (Furtado et al., 2012).
Impact of treatment on children's quality of life | Baseline and 12 months
  The oral health related quality of life will be measured using a validated questionnaire according to the children's age. The "Early Childhood Oral Health Impact Scale" (ECOHIS) (Tesch et al., 2008) will be applied with 4-5 years old patients. The "Child Perceptions Questionnaire" (CPQ) will be used for 6-9 years old patients (Martins et al., 2009). The same questionnaire will be applied immediately before the procedure and on 12 months follow-up. Only one type of questionnaire will be used with each child, according to its age.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade Sao Leopoldo Mandic, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cappiello J. Tratamientos pulpares en incisivos primários. Rev Circ Od Ros 1964;52(4):133-45.
- [Background] de Deus Moura Lde F, de Lima Mde D, Lima CC, Machado JI, de Moura MS, de Carvalho PV. Endodontic Treatment of Primary Molars with Antibiotic Paste: A Report of 38 Cases. J Clin Pediatr Dent. 2016;40(3):175-7. doi: 10.17796/1053-4628-40.3.175. PMID 27472562
- [Background] Furtado GE, Sousa ML, Barbosa TS, Wada RS, Martinez-Mier EA, Almeida ME. [Perceptions of dental fluorosis and evaluation of agreement between parents and children: validation of a questionnaire]. Cad Saude Publica. 2012 Aug;28(8):1493-505. doi: 10.1590/s0102-311x2012000800008. Portuguese. PMID 22892969
- [Background] Guedes-Pinto AC, De Paiva JG, Bozzola JR. [Endodontic treatment of deciduous teeth with pulp necrosis]. Rev Assoc Paul Cir Dent. 1981 May-Jun;35(3):240-4. No abstract available. Portuguese. PMID 6943625
- [Background] Mello-Moura AC, Fanaro J, Nicoletti MA, Mendes FM, Wanderley MT, Guedes-Pinto AC. Variability in the proportion of components of iodoform-based Guedes-Pinto paste mixed by dental students and pediatric dentists. Indian J Dent Res. 2011 Nov-Dec;22(6):781-5. doi: 10.4103/0970-9290.94668. PMID 22484870
- [Background] Monse B, Heinrich-Weltzien R, Benzian H, Holmgren C, van Palenstein Helderman W. PUFA--an index of clinical consequences of untreated dental caries. Community Dent Oral Epidemiol. 2010 Feb;38(1):77-82. doi: 10.1111/j.1600-0528.2009.00514.x. Epub 2009 Dec 7. PMID 20002630
- [Background] Wong DL, Baker CM. Smiling faces as anchor for pain intensity scales. Pain. 2001 Jan;89(2-3):295-300. doi: 10.1016/s0304-3959(00)00375-4. No abstract available. PMID 11291631